CLINICAL TRIAL: NCT06195228
Title: A Retrospective and Prospective Real-world Study of Molecular Typing in the Treatment of Advanced Thyroid Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Shanxi Province Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhejiang Cancer Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Ruijin Hospital (Other); Fujian Cancer Hospital (Other Government); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Shanghai 6th People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai 10th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Changhai Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); The First Affiliated Hospital of Anhui University of Chinese Medicine (Other); Hunan Provincial People's Hospital (Other); Dalian Friendship Hospital Affiliated to Dalian Medical University (Unknown); The Third Affiliated Hospital of Soochow University (Other); Sun Yat-sen University (Other); Liaoning Cancer Hospital & Institute (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associated Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUSCC-TC-RWS01
Record Dates: First submitted 2023-12-23; First posted 2024-01-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Thyroid Cancer Patients Who Received Target Therapy
MeSH Terms: interventions — dabrafenib; trametinib; entrectinib; larotrectinib; pralsetinib; selpercatinib; anlotinib; lenvatinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Radioiodine-refractory differentiated thyroid cancer (Experimental): advanced or metastatic thyroid cancer patients who are refractory to radioiodine treatment
  Interventions: Drug: dabrafenib plus trametinib with or without PD-1 antibody; Drug: entrectinib or larotrectinib with or without anti-PD-1 antibdoy; Drug: pralsetinib or selpercatinib with or without anti-PD-1 antibdoy; Drug: anlotinib or anlotinib plus anti-PD-1 antibody; Drug: lenvatinib plus anti-PD-1 antibody; Drug: Other Targets: precise treatment based on the target
- Differentiated thyroid carcinoma not suitable for radioiodine therapy (Experimental): advanced or metastatic differentiated thyroid cancer patients who are not suitable for radio iodine therapy, for example, DTC patients with huge neck tumor but cannot receive the thyroid ectomy
  Interventions: Drug: dabrafenib plus trametinib with or without PD-1 antibody; Drug: entrectinib or larotrectinib with or without anti-PD-1 antibdoy; Drug: pralsetinib or selpercatinib with or without anti-PD-1 antibdoy; Drug: anlotinib or anlotinib plus anti-PD-1 antibody; Drug: lenvatinib plus anti-PD-1 antibody; Drug: Other Targets: precise treatment based on the target
- Medullary thyroid cancer (Experimental): patients with advanced or metastatic medullary thyroid cancer
  Interventions: Drug: dabrafenib plus trametinib with or without PD-1 antibody; Drug: entrectinib or larotrectinib with or without anti-PD-1 antibdoy; Drug: pralsetinib or selpercatinib with or without anti-PD-1 antibdoy; Drug: anlotinib or anlotinib plus anti-PD-1 antibody; Drug: lenvatinib plus anti-PD-1 antibody; Drug: Other Targets: precise treatment based on the target
- High-grade or poorly differentiated thyroid cancer (Experimental): patients with advanced or metastatic High-grade or poorly differentiated thyroid cancer
  Interventions: Drug: dabrafenib plus trametinib with or without PD-1 antibody; Drug: entrectinib or larotrectinib with or without anti-PD-1 antibdoy; Drug: pralsetinib or selpercatinib with or without anti-PD-1 antibdoy; Drug: anlotinib or anlotinib plus anti-PD-1 antibody; Drug: lenvatinib plus anti-PD-1 antibody; Drug: Other Targets: precise treatment based on the target
- Anaplastic thyroid cancer (Experimental): patients with anaplastic thyroid cancer
  Interventions: Drug: dabrafenib plus trametinib with or without PD-1 antibody; Drug: entrectinib or larotrectinib with or without anti-PD-1 antibdoy; Drug: pralsetinib or selpercatinib with or without anti-PD-1 antibdoy; Drug: anlotinib or anlotinib plus anti-PD-1 antibody; Drug: lenvatinib plus anti-PD-1 antibody; Drug: Other Targets: precise treatment based on the target

INTERVENTIONS:
Drug: dabrafenib plus trametinib with or without PD-1 antibody — advanced thyroid cancer patients who harbor BRAF V600E mutation
Drug: entrectinib or larotrectinib with or without anti-PD-1 antibdoy — advanced thyroid cancer patients who harbor NTRK mutation
Drug: pralsetinib or selpercatinib with or without anti-PD-1 antibdoy — advanced thyroid cancer patients who harbor RET fusion or medullary thyroid carcinoma patients who habor RET mutation.
Drug: anlotinib or anlotinib plus anti-PD-1 antibody — For patients with medullary carcinoma, if there is no RET gene mutation or RET gene mutation is unknown
Drug: lenvatinib plus anti-PD-1 antibody — Advanced thyroid cancer patients who don't harbor the above gene mutation or could not afford the cost of precision treatment even with the above gene mutation
Drug: Other Targets: precise treatment based on the target — Advanced thyroid cancer patients who had other treatment targets not included above

SUMMARY:
This is a retrospective and prospective real-world clinical study of molecular typing in the treatment of advanced thyroid cancer.

The retrospective study : Patients with advanced thyroid cancer who received precise treatment in the 24 participated hospitals from January 2020 to December 2023 were retrieved. The number of previous treatment lines was not limited. Patients who met the inclusion criteria were screened according to the inclusion and exclusion criteria. Demographic information, clinical characteristics, tumor treatment history, medication regimen, adverse reactions, molecular test results, survival follow-up results and other data were collected.

The prospective study : Patients with advanced thyroid cancer who received precise treatment in the 24 Chinese hospitals from January 2024 to April 2027 were enrolled.

DETAILED DESCRIPTION:
see:Arms and Interventions

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent;
2. Each center can be enrolled in patients who meet the age of their own practice range, regardless of gender ;
3. Histologically diagnosed locally advanced or recurrent / metastatic thyroid cancer that cannot undergo radical surgery meets one of the following requirements:

   1. Radioiodine-refractory differentiated thyroid cancer (RAIR-DTC);
   2. Differentiated thyroid carcinoma not suitable for iodine therapy;
   3. Medullary thyroid carcinoma (MTC);
   4. poorly differentiated thyroid cancer (PDTC) or anaplastic thyroid cancer (ATC);
4. Thyroid-related pathogenic or therapeutic target gene detection was performed before enrollment.

Exclusion Criteria:

1. Patients who are participating in clinical trials of other drugs;
2. There is evidence that the patients are pregnant or lactating;
3. Other situations that are not suitable for inclusion in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | up to approximately 3 years
  Complete remission rate+ partial remission rate

SECONDARY OUTCOMES:
Duration of Response(DOR) | up to approximately 3 years
  Time from the date of first partial remission or complete remission to the date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Disease Control Rate(DCR) | up to approximately 3 years
  Complete remission rate+ partial remission rate+stable disease rate
Time to response(TTR) | up to approximately 3 years
  Time from the initiation of the treatment to the first remission
Progression Free Survival(PFS) | up to approximately 3 years
  Time from the date of enrollment to of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Overall survival(OS) | up to approximately 3 years
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, M.D, Principal Investigator — Fudan University; Yu Wang, M.D, Principal Investigator — Fudan University; Qinghai Ji, M.D, Principal Investigator — Fudan University; Yansong Lin, M.D, Principal Investigator — Peking Union Medical College Hospital
Locations (8):
- China (8):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Caixia Liu, Hohhot, Inner Mongolia
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Shanxi, Taiyuan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Peking union medical college hospital, Beijing

IPD SHARING:
Plan to Share IPD: No